CLINICAL TRIAL: NCT07272044
Title: Research on Anesthesia Depth Control Strategy Based on Continuous and Non-invasive Monitoring of Exhaled Breath
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1166
Record Dates: First submitted 2024-06-04; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia
Keywords: Propofol; Breath testing; anesthesia monitoring; Bispectral Index; intravenous and inhalational anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood was analyzed by intraoperative blood gas analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing the first intravenous-inhalation combined anesthesia

SUMMARY:
This study aims to propose a strategy for controlling the depth of anesthesia based on continuous and non-invasive monitoring of exhaled breath: BIS value during intravenous-inhalation combined anesthesia is predicted according to the real-time exhaled concentrations of sevoflurane and propofol, so as to achieve the depth of anesthesia management for patients who cannot use standard BIS. Furthermore, the relationship between anesthetic concentration and depth of anesthesia was analyzed in different subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* ASA I-III
* Expected duration of surgery > 1 hour
* Radial artery catheterization was performed
* Patients requiring BIS monitoring.

Exclusion Criteria:

* Patients with contraindications to general anesthesia
* mental disorder, unable to answer
* long-term use of antiepileptic drugs and psychotropic drugs
* pregnant patients
* patients refused to participate
* the investigator thought that the study was not suitable for inclusion
* patients who did not wake up in PACU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent general anesthesia for the first time and combined intravenous and inhalational anesthesia
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Correlation and consistency analysis between exhaled breath concentrations of two anesthetics and BIS values | 1 day
  Correlation and consistency analysis between exhaled breath concentrations of two anesthetics detected by GC-SAW system and BIS values
Establish a 3D drug dose-effect model of the exhaled concentration and BIS value of anesthetics | 1day
  Establish a 3D drug dose-effect model based on the exhaled gas concentration of anesthetics detected by the GC-SAW system and BIS value

SECONDARY OUTCOMES:
Correlation and consistency analysis of exhaled breath concentration and blood concentration of anesthetics | 1day
  Correlation and consistency analysis of exhaled breath concentration and blood concentration of anesthetics detected by GC-SAW system
The incidence of adverse reactions | 72 hours
  The occurrence of adverse reactions such as postoperative cognitive dysfunction, postoperative nausea and vomiting, chills, and delayed awakening within 72 hours after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China